CLINICAL TRIAL: NCT01203072
Title: A Phase 2b, Randomized, Double-Blind, Multi-Dose Efficacy, Safety and Dose-finding Study of the Oral Factor Xa Inhibitor DU-176b Compared With Placebo for Prevention of Venous Thromboembolism in Patients After Total Knee Arthroplasty (STARS J-1)
Brief Title: A Phase 2b Study of DU-176b, Prevention of Venous Thromboembolism in Patients After Total Knee Arthroplasty
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DU176b-04
Record Dates: First submitted 2010-09-14; First posted 2010-09-16 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2015-01

CONDITIONS: Venous Thromboembolism; Deep Vein Thrombosis; Total Knee Arthroplasty
Keywords: prevention; venous thromboembolism; edoxaban; factor Xa
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis | interventions — edoxaban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- DU-176b 5 mg (Experimental)
  Interventions: Drug: DU-176b
- DU-176b 15 mg (Experimental)
  Interventions: Drug: DU-176b
- DU-176b 30 mg (Experimental)
  Interventions: Drug: DU-176b
- DU-176b 60 mg (Experimental)
  Interventions: Drug: DU-176b
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DU-176b — DU-176b 5mg tablets oral, once daily for 2 weeks
  Other Names: edoxaban
  Arms: DU-176b 5 mg
Drug: DU-176b — DU-176b 15mg tablets, oral once daily for 2 weeks
  Other Names: edoxaban
  Arms: DU-176b 15 mg
Drug: DU-176b — DU-176b 30 mg tablets, oral, once daily for 2 weeks
  Other Names: edoxaban
  Arms: DU-176b 30 mg
Drug: DU-176b — DU-176b 60 mg tablets, oral, once daily for 2 weeks
  Other Names: edoxaban
  Arms: DU-176b 60 mg
Drug: Placebo — Matching placebo oral tablets, once daily for 2 weeks
  Arms: Placebo

SUMMARY:
The objective of this study is to assess the efficacy, safety and dose-response relationship of DU-176b compared with placebo for the prevention of venous thromboembolism in patients after elective total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing unilateral total knee arthroplasty

Exclusion Criteria:

* risks of hemorrhage
* thromboembolic risks
* weight less than 40 kg
* pregnant, suspect pregnancy, or subjects who want to become pregnant

Ages: 20 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 523 (Actual)
Dates: Start 2006-07; Primary Completion 2007-09 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takeshi Fuji, Director, Principal Investigator — Osaka Koseinekin Hospital
Locations (2):
- Japan (2):
  - Osaka
  - Tokyo

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DU-176b 5 mg | DU-176b 15 mg | DU-176b 30 mg | DU-176b 60 mg | Placebo
Started | 105 | 106 | 104 | 106 | 102
Completed | 95 | 100 | 101 | 100 | 96
Not Completed | 10 | 6 | 3 | 6 | 6
Not completed — Adverse Event | 5 | 3 | 2 | 4 | 2
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 2 | 1 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DU-176b 5 mg | DU-176b 15 mg | DU-176b 30 mg | DU-176b 60 mg | Placebo | Total
Number analyzed (Participants) | 88 | 92 | 88 | 88 | 89 | 445
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.2 (7.7) | 71.7 (7.0) | 71.6 (8.1) | 72.1 (7.0) | 70.3 (6.5) | 71.2 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 74 | 69 | 69 | 68 | 347
  Male | 21 | 18 | 19 | 19 | 21 | 98
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 88 | 92 | 88 | 88 | 89 | 445
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 88 | 92 | 88 | 88 | 89 | 445

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With Venous Thromboembolism Events.
Description: The primary efficacy endpoint was the proportion of subjects who experienced at least one of the thromboembolic events listed below during the period from the start of study treatment to the venography at the end of study treatment.
  * Lower extremity DVT confirmed by bilateral venography at the end of study treatment
  * Definite diagnosis of symptomatic PE
  * Symptomatic DVT confirmed before the venography at the end of study treatment The objectives were to verify the non-inferiority of edoxaban to enoxaparin with regard to prevention of VTE
Time Frame: 2 weeks
Population: The FAS was defined as all subjects enrolled in the study, but excluded those who had significant GCP violations, who had not received any doses of the study drug, or those who did not develop symptomatic DVT or PE, but in whom venography was not appropriately performed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | DU-176b 5 mg | DU-176b 15 mg | DU-176b 30 mg | DU-176b 60 mg | Placebo
Number analyzed (Participants) | 88 | 92 | 88 | 88 | 89
percentage of participants | 29.5 [20.0 to 39.1] | 26.1 [17.1 to 35.1] | 12.5 [5.6 to 19.4] | 9.1 [3.1 to 15.1] | 48.3 [37.9 to 58.7]
Statistical Analysis 1: Comparison: DU-176b 5 mg vs DU-176b 15 mg vs DU-176b 30 mg vs DU-176b 60 mg vs Placebo; As the primary analysis, the dose-response relationship in the incidence of thromboembolic event was verified using the Cochran-Armitage test; Test type: Superiority or Other; p < 0.001, Cochran-Armitage — Significance level for Cochran-Armitage test and comparison using Shirley-Williams method was set at one-sided, 0.025. For other tests, significance level and confidence coefficient were set at two-sided, 0.05 and 0.95, respectively, unless specified

2. Secondary Outcome: Incidence of Major Bleeding or Clinically Relevant Non-major Bleeding
Description: Incidence of Major Bleeding or Clinically Relevant Non-major Bleeding. Related to the study drug
Time Frame: 2 weeks
Population: Safety Analysis Set is defined as subjects secondarily enrolled in study, but excluded those with significant GCP violations, did not receive any doses of study drug, or had no safety data after start of study treatment. Subjects with significant GCP violations, but received at least one dose of study drug, safety data were assessed individually
Measure: Number (95% Confidence Interval); unit: percentage of subjects with bleeds
Arm/Group | DU-176b 5 mg | DU-176b 15 mg | DU-176b 30 mg | DU-176b 60 mg | Placebo
Number analyzed (Participants) | 103 | 106 | 103 | 106 | 102
percentage of subjects with bleeds | 1.9 [0.5 to 6.8] | 3.8 [1.5 to 9.3] | 3.9 [1.5 to 9.6] | 4.7 [2.0 to 10.6] | 3.9 [1.5 to 9.7]

ADVERSE EVENTS:
Arm/Group | DU-176b 5 mg | DU-176b 15 mg | DU-176b 30 mg | DU-176b 60 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 2/103 | 1/106 | 1/103 | 3/106 | 5/102
Other Adverse Events (participants affected / at risk) | 78/103 | 85/106 | 78/103 | 78/106 | 67/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DU-176b 5 mg (N=103) | DU-176b 15 mg (N=106) | DU-176b 30 mg (N=103) | DU-176b 60 mg (N=106) | Placebo (N=102)
nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DU-176b 5 mg (N=103) | DU-176b 15 mg (N=106) | DU-176b 30 mg (N=103) | DU-176b 60 mg (N=106) | Placebo (N=102)
nasopharyngitis (Infections and infestations) | 7 (7) | 9 (9) | 10 (10) | 4 (4) | 8 (8)
insomnia (Psychiatric disorders) | 2 (2) | 4 (4) | 8 (9) | 4 (4) | 5 (5)
headache (Nervous system disorders) | 1 (1) | 5 (5) | 6 (6) | 2 (2) | 4 (4)
wound haemorrhage (Vascular disorders) | 3 (3) | 2 (2) | 1 (1) | 6 (7) | 0 (0)
constipation (Gastrointestinal disorders) | 5 (5) | 6 (6) | 4 (4) | 4 (4) | 5 (5)
diarrhea (Gastrointestinal disorders) | 7 (7) | 3 (3) | 5 (5) | 4 (4) | 7 (8)
dermatitis contact (Skin and subcutaneous tissue disorders) | 4 (4) | 7 (7) | 2 (2) | 2 (2) | 1 (1)
erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 6 (6) | 3 (3) | 2 (2)
heamorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4) | 7 (7) | 5 (5) | 4 (4)
pruritis (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (6) | 6 (8) | 1 (1) | 1 (1)
haematuria (Renal and urinary disorders) | 2 (2) | 4 (4) | 1 (1) | 7 (8) | 0 (0)
alanine aminotransferase increased (Investigations) | 7 (7) | 7 (7) | 7 (7) | 6 (6) | 8 (9)
aspartate aminotransferase increased (Investigations) | 7 (7) | 7 (7) | 7 (7) | 4 (4) | 6 (6)
blood lactate dehydrogenase increased (Investigations) | 13 (13) | 17 (17) | 16 (16) | 16 (17) | 12 (12)
gamma glutamyltransferase increased (Investigations) | 10 (10) | 10 (10) | 7 (7) | 11 (11) | 7 (7)
blood urine present (Investigations) | 6 (6) | 9 (10) | 9 (10) | 15 (16) | 6 (7)
haemoglobin decreased (Investigations) | 3 (3) | 6 (6) | 6 (6) | 7 (7) | 5 (5)
platelet count increased (Investigations) | 9 (9) | 14 (14) | 12 (12) | 6 (6) | 5 (5)
blood alkaline phosphate increased (Investigations) | 11 (11) | 12 (12) | 9 (9) | 11 (11) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall not publish the results of the Study at any time without the prior written approval of Sponsor.